CLINICAL TRIAL: NCT00857844
Title: Genetic Predisposition of Chronic Nephrotoxicity From Calcineurin Inhibitors in Liver Transplant Recipients, Potential Correlation With Urinary Biomarkers
Brief Title: Genetic Predisposition-Chronic Nephrotoxicity From CI-Liver Transplant Recipients-Potential Correlation-Urinary Biomarkers
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Gallon, Associate Professor, Northwestern University
Other Study IDs: STU8309 0773-018
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Complication of Transplanted Liver
Keywords: Chronic Nephrotoxicity; Kidney dysfunction post liver transplant; Urinary biomarkers of chronic nephrotoxicity from CI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Urine will be collected from all patients in the 3 groups and analyzed for biomarkers of interstitial fibrosis and proximal tubule injury. Specific biomarkers that will be tested are: urinary TGF-beta1, kidney injury molecule-1 and angiotensinogen. Urinary biomarkers will be normalized to creatinine and analyzed using an ELISA assay.
  * An additional 18mls of blood will be collected. This blood will be used to study organ transplant tolerance in subjects who are currently using immunosuppressant medications.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Normal GFR (>90ml/min/1.73m2). Stage I CKD
- Group 2: GFR between 30-59ml/min/1.73m2. Stage III CKD
- Group 3: GFR between 15-29ml/min/1.72m2. Stage IV CKD

SUMMARY:
The purpose of this study is to determine the relationship between genomic variants of components of the renin-angiotensin system and the development of kidney problems due to Calcineurin-inhibitors post liver transplant.Also the investigator will evaluate the relationship between chronic renal failure post liver transplant and the risk of death. A sample of blood and urine wil be examined to see how the patient's genes are arranged in order to determine the difference in genes between people which may explain who will develop chronic renal failure after having received a liver transplant.

The results may help us classify patients according to their risk and allow us to target their treatment to their individual need. In addition, it may ultimately lead to treatments that slows or prevents the development of chronic rejection.

DETAILED DESCRIPTION:
Study Design:

This study will be a cross-sectional investigation of liver transplant recipients who received a liver transplant and have at least 6 months of follow-up. This study will be conducted at Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation and Northwestern University.

Patients who underwent liver transplantation and have at least 6 months of follow-up receiving a maintenance immunosuppression (which consists of calcineurin inhibitors (CI), cyclosporine (CsA), or tacrolimus (Tac)) during the entire post-transplant follow-up period will be included in the analysis.

For each patient, the following information will be collected:

* Date of transplantation, age, gender, race, causes of liver failure, past medical history including incidence of hypertension, diabetes mellitus, post-operative complications, post-operative infections, number of acute liver rejection episodes, death, CsA and Tac trough levels at different time points post-transplant and sCr levels before liver transplant, at 1, 6, 12, 24 months, and yearly post-transplant.
* GFR (Glomerular Filtration Rate) with MDRD equation before liver transplant, at 1, 6, 12, 24 months, and yearly post-transplant.
* In the attempt to rule out all patients with pre-existing CRF before liver transplant, only the patients with sCr<1.0mg/dL before liver transplant will be included in our analysis.

Genotyping:

* DNA will be extracted using blood buffy coat from liver transplant recipients.
* Determination of ACE genotypes will be performed by using polymerase chain reaction sequence-specific primers (PCR-SSP) and polymerase chain reaction restriction fragment length polymorphism (PCR-RFLP).
* Based on GRF calculation by MDRD equation liver transplant patients will be categorized into three groups based on NKF staging of chronic kidney disease:

Group I->normal GFR (>90ml/min/1.73m2). Stage I CKD Group II->GFR between 30-59ml/min/1.73m2. Stage III CKD Group III->GFR between 15-29ml/min/1.72m2. Stage IV CKD

* Urine (80cc) will be collected from all patients in the 3 groups and analyzed for biomarkers of interstitial fibrosis and proximal tubule injury. Specific biomarkers that will be tested are: urinary TGF-beta1, kidney injury molecule-1 and angiotensinogen. Urinary biomarkers will be normalized to creatinine and analyzed using an ELISA assay.
* Blood (20cc)will be taken at one visit.
* An additional blood draw (18cc) will be requested from all subjects. This blood will be used to study organ transplant tolerance in subjects who are currently using immunosuppressant medications.

Statistical Plan-Statistical tests to be performed:

Once liver transplant patients are genotyped and urine samples are collected we will compared the development of CKD post liver transplant for associations with urinary biomarkers and polymorphisms of the ACE gene. Two sample t tests will be used to compare differences in continuous variables between liver patients with different degree of CKD; chi square tests will be used to compare differences in discrete variables. Multivariable logistic regression analysis will be also performed to identify the combination of clinical variable and gene polymorphisms that are significantly associated with the development of post liver transplant renal dysfunction.

This study will enable us to learn and evaluate potential genetic predisposition for the development of renal dysfunction after exposure to CI. If our hypothesis is correct, testing of the component of the RAS genotypes may help identify patients at risk for CI nephrotoxicity and help in the pre-selection of liver transplant candidates in whom the use of CI as primary immunosuppression should be avoided.

Furthermore, the data generated from this study might serve as a strong basis for a prospective NIH-founded project to look at the role of agents that block the renin-angiotensin system for the prevention of CI-induced chronic nephrotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Males and females > 18 years old
* Liver transplant recipients who have received a liver transplant at least 6 months ago
* Liver transplant recipients receiving a maintenance immunosuppression.

Exclusion Criteria:

* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the study
* Pre-existing known kidney disease before liver transplantation
* Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in liver transplant recipients. We are planning to collect data and genotyping in 650 liver transplant recipients. Patients who satisfy the following inclusion/exclusion criteria will be eligible for the study:
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To investigate, in liver transplant patients, the role of urinary biomarkers as indirect indices of chronic nephrotoxicity from CI and associate, where possible, urinary biomarkers to genomic variants of the angiotensin converting | At time of enrollment
  Blood draw (20cc) and urine collection (80cc).

SECONDARY OUTCOMES:
The study will also evaluate if specific demographic characteristics are associated with an increased risk of nephrotoxic damage from CI. | At time of enrollment
  Blood draw (20cc)
Organ transplant tolerance in subjects who are currently using immunosuppressant medications. | One additional blood draw - follow-up time point
  Blood draw (18cc).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, M.D., Principal Investigator — Northwestern University, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Bennett WM. Insights into chronic cyclosporine nephrotoxicity. Int J Clin Pharmacol Ther. 1996 Nov;34(11):515-9. PMID 8937936
- [Background] Bennett WM, DeMattos A, Meyer MM, Andoh T, Barry JM. Chronic cyclosporine nephropathy: the Achilles' heel of immunosuppressive therapy. Kidney Int. 1996 Oct;50(4):1089-100. doi: 10.1038/ki.1996.415. No abstract available. PMID 8887265
- [Background] Myers BD. Cyclosporine nephrotoxicity. Kidney Int. 1986 Dec;30(6):964-74. doi: 10.1038/ki.1986.280. No abstract available. PMID 3546916
- [Background] Puschett JB, Greenberg A, Holley J, McCauley J. The spectrum of ciclosporin nephrotoxicity. Am J Nephrol. 1990;10(4):296-309. doi: 10.1159/000168123. No abstract available. PMID 2240057
- [Background] Young EW, Ellis CN, Messana JM, Johnson KJ, Leichtman AB, Mihatsch MJ, Hamilton TA, Groisser DS, Fradin MS, Voorhees JJ. A prospective study of renal structure and function in psoriasis patients treated with cyclosporin. Kidney Int. 1994 Oct;46(4):1216-22. doi: 10.1038/ki.1994.387. PMID 7861719
- [Background] Myers BD, Ross J, Newton L, Luetscher J, Perlroth M. Cyclosporine-associated chronic nephropathy. N Engl J Med. 1984 Sep 13;311(11):699-705. doi: 10.1056/NEJM198409133111103. PMID 6382005
- [Background] Goldstein DJ, Zuech N, Sehgal V, Weinberg AD, Drusin R, Cohen D. Cyclosporine-associated end-stage nephropathy after cardiac transplantation: incidence and progression. Transplantation. 1997 Mar 15;63(5):664-8. doi: 10.1097/00007890-199703150-00009. PMID 9075835
- [Background] Hornberger J, Best J, Geppert J, McClellan M. Risks and costs of end-stage renal disease after heart transplantation. Transplantation. 1998 Dec 27;66(12):1763-70. doi: 10.1097/00007890-199812270-00034. PMID 9884274
- [Background] Fisher NC, Nightingale PG, Gunson BK, Lipkin GW, Neuberger JM. Chronic renal failure following liver transplantation: a retrospective analysis. Transplantation. 1998 Jul 15;66(1):59-66. doi: 10.1097/00007890-199807150-00010. PMID 9679823
- [Background] Gonwa TA, Mai ML, Melton LB, Hays SR, Goldstein RM, Levy MF, Klintmalm GB. End-stage renal disease (ESRD) after orthotopic liver transplantation (OLTX) using calcineurin-based immunotherapy: risk of development and treatment. Transplantation. 2001 Dec 27;72(12):1934-9. doi: 10.1097/00007890-200112270-00012. PMID 11773892
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Mervaala E, Lassila M, Vaskonen T, Krogerus L, Lahteenmaki T, Vapaatalo H, Karppanen H. Effects of ACE inhibition on cyclosporine A-induced hypertension and nephrotoxicity in spontaneously hypertensive rats on a high-sodium diet. Blood Press. 1999;8(1):49-56. doi: 10.1080/080370599438392. PMID 10412883
- [Background] Perico N, Benigni A, Bosco E, Rossini M, Orisio S, Ghilardi F, Piccinelli A, Remuzzi G. Acute cyclosporine A nephrotoxicity in rats: which role for renin-angiotensin system and glomerular prostaglandins? Clin Nephrol. 1986;25 Suppl 1:S83-8. PMID 3519031
- [Background] Shihab FS, Bennett WM, Tanner AM, Andoh TF. Angiotensin II blockade decreases TGF-beta1 and matrix proteins in cyclosporine nephropathy. Kidney Int. 1997 Sep;52(3):660-73. doi: 10.1038/ki.1997.380. PMID 9291185
- [Background] Pichler RH, Franceschini N, Young BA, Hugo C, Andoh TF, Burdmann EA, Shankland SJ, Alpers CE, Bennett WM, Couser WG, et al. Pathogenesis of cyclosporine nephropathy: roles of angiotensin II and osteopontin. J Am Soc Nephrol. 1995 Oct;6(4):1186-96. doi: 10.1681/ASN.V641186. PMID 8589285
- [Background] Burdmann EA, Andoh TF, Yu L, Bennett WM. Cyclosporine nephrotoxicity. Semin Nephrol. 2003 Sep;23(5):465-76. doi: 10.1016/s0270-9295(03)00090-1. PMID 13680536
- [Background] Feria I, Pichardo I, Juarez P, Ramirez V, Gonzalez MA, Uribe N, Garcia-Torres R, Lopez-Casillas F, Gamba G, Bobadilla NA. Therapeutic benefit of spironolactone in experimental chronic cyclosporine A nephrotoxicity. Kidney Int. 2003 Jan;63(1):43-52. doi: 10.1046/j.1523-1755.2003.00707.x. PMID 12472767
- [Background] Beohar N, Damaraju S, Prather A, Yu QT, Raizner A, Kleiman NS, Roberts R, Marian AJ. Angiotensin-I converting enzyme genotype DD is a risk factor for coronary artery disease. J Investig Med. 1995 Jun;43(3):275-80. PMID 7614074
- [Background] Rigat B, Hubert C, Alhenc-Gelas F, Cambien F, Corvol P, Soubrier F. An insertion/deletion polymorphism in the angiotensin I-converting enzyme gene accounting for half the variance of serum enzyme levels. J Clin Invest. 1990 Oct;86(4):1343-6. doi: 10.1172/JCI114844. PMID 1976655
- [Background] Hingorani AD, Brown MJ. A simple molecular assay for the C1166 variant of the angiotensin II type 1 receptor gene. Biochem Biophys Res Commun. 1995 Aug 15;213(2):725-9. doi: 10.1006/bbrc.1995.2190. PMID 7646529
- [Background] Lindpaintner K, Pfeffer MA, Kreutz R, Stampfer MJ, Grodstein F, LaMotte F, Buring J, Hennekens CH. A prospective evaluation of an angiotensin-converting-enzyme gene polymorphism and the risk of ischemic heart disease. N Engl J Med. 1995 Mar 16;332(11):706-11. doi: 10.1056/NEJM199503163321103. PMID 7854377
- [Background] Morris BJ, Monaghan JC, Perich R, Stokes GS, Jackson B, Schrader AP. Genotypic influence on plasma dipeptidyl carboxypeptidase-1 activity in hypertensives. Clin Exp Pharmacol Physiol. 1994 Apr;21(4):343-6. doi: 10.1111/j.1440-1681.1994.tb02525.x. PMID 7923904
- [Background] Danser AH, Schalekamp MA, Bax WA, van den Brink AM, Saxena PR, Riegger GA, Schunkert H. Angiotensin-converting enzyme in the human heart. Effect of the deletion/insertion polymorphism. Circulation. 1995 Sep 15;92(6):1387-8. doi: 10.1161/01.cir.92.6.1387. PMID 7664416
- [Background] Inoue I, Nakajima T, Williams CS, Quackenbush J, Puryear R, Powers M, Cheng T, Ludwig EH, Sharma AM, Hata A, Jeunemaitre X, Lalouel JM. A nucleotide substitution in the promoter of human angiotensinogen is associated with essential hypertension and affects basal transcription in vitro. J Clin Invest. 1997 Apr 1;99(7):1786-97. doi: 10.1172/JCI119343. PMID 9120024
- [Background] Jeunemaitre X, Inoue I, Williams C, Charru A, Tichet J, Powers M, Sharma AM, Gimenez-Roqueplo AP, Hata A, Corvol P, Lalouel JM. Haplotypes of angiotensinogen in essential hypertension. Am J Hum Genet. 1997 Jun;60(6):1448-60. doi: 10.1086/515452. PMID 9199566
- [Background] Vleming LJ, van der Pijl JW, Lemkes HH, Westendorp RG, Maassen JA, Daha MR, van Es LA, van Kooten C. The DD genotype of the ACE gene polymorphism is associated with progression of diabetic nephropathy to end stage renal failure in IDDM. Clin Nephrol. 1999 Mar;51(3):133-40. PMID 10099885
- [Background] Harden PN, Geddes C, Rowe PA, McIlroy JH, Boulton-Jones M, Rodger RS, Junor BJ, Briggs JD, Connell JM, Jardine AG. Polymorphisms in angiotensin-converting-enzyme gene and progression of IgA nephropathy. Lancet. 1995 Jun 17;345(8964):1540-2. doi: 10.1016/s0140-6736(95)91088-3. PMID 7791440
- [Background] van Essen GG, Rensma PL, de Zeeuw D, Sluiter WJ, Scheffer H, Apperloo AJ, de Jong PE. Association between angiotensin-converting-enzyme gene polymorphism and failure of renoprotective therapy. Lancet. 1996 Jan 13;347(8994):94-5. doi: 10.1016/s0140-6736(96)90213-5. PMID 8538349
- [Background] Broekroelofs J, Stegeman CA, Navis G, Tegzess AM, De Zeeuw D, De Jong PE. Risk factors for long-term renal survival after renal transplantation: a role for angiotensin-converting enzyme (insertion/deletion) polymorphism? J Am Soc Nephrol. 1998 Nov;9(11):2075-81. doi: 10.1681/ASN.V9112075. PMID 9808093
- [Background] Barocci S, Ginevri F, Valente U, Torre F, Gusmano R, Nocera A. Correlation between angiotensin-converting enzyme gene insertion/deletion polymorphism and kidney graft long-term outcome in pediatric recipients: a single-center analysis. Transplantation. 1999 Feb 27;67(4):534-8. doi: 10.1097/00007890-199902270-00008. PMID 10071023
- [Background] Gallon L, Akalin E, Lynch P, Rothberg L, Parker M, Schiano T, Abecassis M, Murphy B. ACE gene D/D genotype as a risk factor for chronic nephrotoxicity from calcineurin inhibitors in liver transplant recipients. Transplantation. 2006 Feb 15;81(3):463-8. doi: 10.1097/01.tp.0000185305.63759.d3. PMID 16477235
- [Background] Han WK, Bailly V, Abichandani R, Thadhani R, Bonventre JV. Kidney Injury Molecule-1 (KIM-1): a novel biomarker for human renal proximal tubule injury. Kidney Int. 2002 Jul;62(1):237-44. doi: 10.1046/j.1523-1755.2002.00433.x. PMID 12081583
- [Background] Parikh CR, Jani A, Mishra J, Ma Q, Kelly C, Barasch J, Edelstein CL, Devarajan P. Urine NGAL and IL-18 are predictive biomarkers for delayed graft function following kidney transplantation. Am J Transplant. 2006 Jul;6(7):1639-45. doi: 10.1111/j.1600-6143.2006.01352.x. PMID 16827865
- [Background] Amer H, Lieske J, Grande J, Stegall M, Larson T. Urinary TGF-beta1 predicts progressive renal allograft fibrosis on one year protocol biopsies. Abstract, ASN, 2006. San Diego
- [Background] Iwazu Y, Muto S, Hirahara I, Fujisawa G, Miyata Y, Kusano E. Urinary matrix metalloproteinase is a useful marker for the development of Deoxycorticosterone Acetate/salt-induced tubulointerstitial fibrosis. Abstract, ASN, 2006. San Diego
- [Background] van Timmeren MM, van den Heuvel MC, Bailly V, Bakker SJ, van Goor H, Stegeman CA. Tubular kidney injury molecule-1 (KIM-1) in human renal disease. J Pathol. 2007 Jun;212(2):209-17. doi: 10.1002/path.2175. PMID 17471468
- [Background] Yamamoto T, Nakagawa T, Suzuki H, Ohashi N, Fukasawa H, Fujigaki Y, Kato A, Nakamura Y, Suzuki F, Hishida A. Urinary angiotensinogen as a marker of intrarenal angiotensin II activity associated with deterioration of renal function in patients with chronic kidney disease. J Am Soc Nephrol. 2007 May;18(5):1558-65. doi: 10.1681/ASN.2006060554. Epub 2007 Apr 4. PMID 17409316